CLINICAL TRIAL: NCT02221011
Title: The Effect of Extracorporeal Shock Wave Therapy on Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGHIRB: 2-102-05-018
Record Dates: First submitted 2014-08-14; First posted 2014-08-20 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Spasticity
Keywords: Shock wave; Spasticity; Effect
MeSH Terms: conditions — Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- shock wave (three times) (Experimental): E-SWT, Elettronica Pagani, Italy 3.5 bars 1500 beats in FCU, FCR 3 bars 4000 beats diffuse in intrinsic muscle Once a week for 3 weeks
  Interventions: Device: Shock wave
- Sham shock wave (Sham Comparator): E-SWT, Elettronica Pagani, Italy Sham without energy, 1500 beats in FCU, FCR and 4000 beats diffuse in intrinsic muscle
  Interventions: Device: Shock wave
- Shock wave (one time) (Experimental): E-SWT, Elettronica Pagani, Italy 3.5 bars 1500 beats in FCU, FCR 3 bars 4000 beats diffuse in intrinsic muscle Only one dose
  Interventions: Device: Shock wave

INTERVENTIONS:
Device: Shock wave — Shock waves are defined a sequence of acoustic pulse characterized by a high peak pressure (100 MPa), fast pressure rise (< 10 ns) and short duration (10 μs) is conveyed by an appropriate generator to a specific target area with an energy density in the range of 0.003-0.890 mJ/mm2.
  Different studies and clinical experiments have demonstrated the efficacy of shock waves in the treatment of musculoskeletal system such as chronic tendinopathies, calcific tendinitis of the shoulder, lateral epicondylitis, plantar fasciitis, and several tendon diseases.
  Other Names: E-SWT

SUMMARY:
The effect of traditional treatment for spasticity is barely satisfactory. The shock wave has been used to treat the spasticity with expressively response and the effect could persist for 1-3 months in different studies. However most sutdies lack the sham or control group. The purpose of this study was to assess the effect of shock wave for spasticity in wrist and hand.

DETAILED DESCRIPTION:
The patients with spasticity for at least 6 months were randomized for 3 groups. Group I: patients receive one session of shock wave per week for 3 weeks; Group II: patients receive only one session of shock wave; Group III: patients receive the sham shock wave per week for 3 weeks. The outcome measurements include Modified Asthow scale, passive range of motion, Disability Assessment Scale and Fugl-Meyer Assessment Scale (hand function and wrist control).

ELIGIBILITY:
Inclusion Criteria:

Age between 20-80 year-old Spasticity measured as Modified Asthow Scale more than 1+ point and persist at least 6 months Clear consciousness No receive Phenol injection or Botulinum toxin in past 6 months

Exclusion Criteria:

Cancer Joint contracture Coagulopathy Pregnancy Pacemaker Inflammation status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of spasticity on 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment.
  Using the modyfied Ashworth Scale to measure the spasticity before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline of range of motion on 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment.
  Using the digital goniometer to measure the passive range of motion before treatment and multiple time frame after treatment.
Change from baseline of pain on 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment.
  Using the Visual analog scale (VAS) to measure the pain from spasticity scale before treatment and multiple time frame after treatment.
Change from baseline of disability on 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment.
  Using the Disability Assessment Scale to measure the disabilty scale before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Tri-Service General Hospital National Defense Medical Center
Locations (1):
- Tri-Service General Hospital National Defense Medical Center, Taipei, Neihu, Taiwan

REFERENCES:
- [Background] Rompe JD, Hope C, Kullmer K, Heine J, Burger R. Analgesic effect of extracorporeal shock-wave therapy on chronic tennis elbow. J Bone Joint Surg Br. 1996 Mar;78(2):233-7. PMID 8666632
- [Background] Loew M, Daecke W, Kusnierczak D, Rahmanzadeh M, Ewerbeck V. Shock-wave therapy is effective for chronic calcifying tendinitis of the shoulder. J Bone Joint Surg Br. 1999 Sep;81(5):863-7. doi: 10.1302/0301-620x.81b5.9374. PMID 10530851
- [Background] Manganotti P, Amelio E. Long-term effect of shock wave therapy on upper limb hypertonia in patients affected by stroke. Stroke. 2005 Sep;36(9):1967-71. doi: 10.1161/01.STR.0000177880.06663.5c. Epub 2005 Aug 18. PMID 16109905
- [Background] Vidal X, Morral A, Costa L, Tur M. Radial extracorporeal shock wave therapy (rESWT) in the treatment of spasticity in cerebral palsy: a randomized, placebo-controlled clinical trial. NeuroRehabilitation. 2011;29(4):413-9. doi: 10.3233/NRE-2011-0720. PMID 22207070
- [Background] Sohn MK, Cho KH, Kim YJ, Hwang SL. Spasticity and electrophysiologic changes after extracorporeal shock wave therapy on gastrocnemius. Ann Rehabil Med. 2011 Oct;35(5):599-604. doi: 10.5535/arm.2011.35.5.599. Epub 2011 Oct 31. PMID 22506181